CLINICAL TRIAL: NCT04294472
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Pharmacokinetics and Efficacy of MAU868 for the Treatment of BK Viremia in Kidney Transplant Recipients (Neutra4)
Brief Title: A Safety, Pharmacokinetics and Efficacy Study of MAU868 for the Treatment of BK Viremia in Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAU868-201
Record Dates: First submitted 2020-02-26; First posted 2020-03-04 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-02

CONDITIONS: BK Virus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1: MAU868 1350 mg IV approximately every 28 days for a total of 4 doses
  Interventions: Drug: MAU868
- Cohort 2 (Experimental): Cohort 2: MAU868 6750 mg IV on Study Day 1 and then 1350 mg IV approximately every 28 days for a total of 4 doses
  Interventions: Drug: MAU868
- Cohort 3 (Experimental): Cohort 3: MAU868 6750 mg IV approximately every 28 days for a total of 4 doses
  Interventions: Drug: MAU868
- Placebo Cohort 1, 2, 3 (Placebo Comparator): 5% dextrose in water [D5W] IV delivered every 28 days for a total of 4 doses
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MAU868 — MAU868 is a human monoclonal antibody (IgG1) that binds the viral capsid protein, VP1, that is responsible for binding to the surface of host cells
  Arms: Cohort 1; Cohort 2; Cohort 3
Other: Placebo — 250 mL D5W placebo IV to be labeled to match that of MAU868
  Arms: Placebo Cohort 1, 2, 3

SUMMARY:
This clinical research study will test the safety and efficacy of the investigational medication MAU868, compared to a placebo, in patients who have had a kidney transplant who have active BK virus.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female 18 years of age or older.
* Recipient of a kidney (or kidney-pancreas) transplant within the year prior to enrollment
* Documented BKV viremia based on local or central laboratory testing within 10 days

Exclusion Criteria:

* A BKV plasma viral load which has exceeded 10^3 copies/mL for >4 months.
* A BKV plasma viral load of ≥ 10^7 copies/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - University of Kentucky, Lexington, Kentucky
  - The Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Renal Disease Research Institute, LLC, Dallas, Texas
  - The University of Texas Southwester Medical Center, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - University of Washington, Seattle, Washington
- Canada (3):
  - University Health Network, Toronto, Ontario
  - Centre intégré universitaire de santé et de services sociaux (CIUSSS) de l'Est de-l'Île-de-Montréal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Helle F, Aubry A, Morel V, Descamps V, Demey B, Brochot E. Neutralizing Antibodies Targeting BK Polyomavirus: Clinical Importance and Therapeutic Potential for Kidney Transplant Recipients. J Am Soc Nephrol. 2024 Oct 1;35(10):1425-1433. doi: 10.1681/ASN.0000000000000457. Epub 2024 Jul 9. PMID 39352862

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: 5% dextrose in water [D5W] IV delivered every 28 days for a total of 4 doses
- Active Arm (Cohort 1): MAU868 1350 mg every 28 days for a total of 4 doses
- Active Arm (Cohort 2): MAU868 6750 once and 1350 mg every 28 days for a total of 4 doses
Period: Overall Study
Arm/Group | Placebo | Active Arm (Cohort 1) | Active Arm (Cohort 2)
Started | 8 | 11 | 11
Completed | 8 | 9 | 9
Not Completed | 0 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Randomized but not treated | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Participant Flow module included 30 participants randomized; two subjects randomized but not treated were identified, leaving 28 randomized and treated subjects in subsequent modified intent-to-treat analyses. Overall Number of Baseline Participants was based on 28 randomized and treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Arm (Cohort 1) | Active Arm (Cohort 2) | Total
Number analyzed (Participants) | 8 | 10 | 10 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 8 | 20
  >=65 years | 2 | 4 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (16.85) | 60.1 (13.52) | 56.2 (8.50) | 56.5 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 5 | 9 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 5
  Not Hispanic or Latino | 8 | 7 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 1 | 9
  White | 3 | 4 | 7 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 2 | 3
  United States | 8 | 9 | 8 | 25
eGFR (CK-EPI)(mL/min/ 1.73m^2) [Mean (Standard Deviation); unit: mL/min/ 1.73m^2] | 59.5 (21.23) | 54.1 (22.93) | 51.1 (11.53) | 54.6 (18.66)
Time from Kidney Transplant (days) [Mean (Standard Deviation); unit: Days] | 174.6 (82.57) | 175.6 (93.53) | 143.5 (89.72) | 163.9 (87.21)
Baseline Plasma Viral Load (copies/mL) based on central lab [Mean (Standard Deviation); unit: copies/mL] | 315100.0 (620601.58) | 85100.0 (152159.91) | 24690.0 (36203.73) | 129239.3 (350731.32)
Duration of BK Viremia (days) [Mean (Standard Deviation); unit: Days] | 58.4 (23.11) | 56.6 (39.33) | 41.9 (23.74) | 51.9 (29.99)

OUTCOME MEASURES:

1. Primary Outcome: Time (Weeks) to Decrease of BKV Plasma Viral Load by 1 Log
Description: The efficacy of MAU868 in treating BK viremia will be measured primarily by measuring the BK Viral Load in the plasma over time.
Time Frame: Study Week 1 - Study Week 36
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Active Arm (Cohort 1) | Active Arm (Cohort 2)
Number analyzed (Participants) | 8 | 10 | 10
Weeks | 19.61 (11.75) | 10.80 (11.50) | 18.25 (16.28)
Statistical Analysis 1: Comparison: Placebo vs Active Arm (Cohort 1); Test type: Superiority — Cohort 1 vs Placebo; p = 0.1866, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Active Arm (Cohort 2); Test type: Superiority — Cohort 2 vs Placebo; p = 0.2627, Log Rank

2. Primary Outcome: Time (Weeks) to First Decrease of BKV Plasma Viral Load to Less Than Lower Limit of Quantification (LLOQ)
Description: as for outcome 1
Time Frame: Study Week 1 - Study Week 36
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Active Arm (Cohort 1) | Active Arm (Cohort 2)
Number analyzed (Participants) | 8 | 10 | 10
Weeks | NA (NA) — No subjects in placebo group achieved BKV plasma viral load to less than lower limit of quantification | 16.79 (13.57) | 8.18 (6.46)
Statistical Analysis 1: Comparison: Placebo vs Active Arm (Cohort 1); Test type: Superiority — Cohort 1 vs Placebo; p = 0.0639, Log Rank
Statistical Analysis 2: Comparison: Placebo vs Active Arm (Cohort 2); Test type: Superiority — Cohort 2 vs Placebo; p = 0.0508, Log Rank

ADVERSE EVENTS:
Time Frame: Study Week 1 - Study Week 36
Description: The Participant Flow module included 30 participants randomized; two subjects randomized but not treated were identified, leaving 28 randomized and treated subjects in subsequent modified intent-to-treat analyses. The Total Number of Participants at Risk was based on 28 randomized and treated participants.
Arm/Group | Placebo | Active Arm (Cohort 1) | Active Arm (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/8 | 1/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 2/8 | 6/10 | 6/10
Other Adverse Events (participants affected / at risk) | 8/8 | 9/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Active Arm (Cohort 1) (N=10) | Active Arm (Cohort 2) (N=10)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Active Arm (Cohort 1) (N=10) | Active Arm (Cohort 2) (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic allograft nephropathy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BK virus infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (5)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 1 (3)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT04294472/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT04294472/SAP_001.pdf